CLINICAL TRIAL: NCT01821443
Title: A Single Arm Study of Neurocognitive Outcomes in Patients With Brain Metastases Managed Primarily With Stereotactic Radiosurgery (SRS)
Brief Title: A Single Arm Study of Neurocognitive Outcomes in Patients With Brain Metastases Managed With Stereotactic Radiosurgery (SRS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: University of California, San Francisco (Other)
Collaborators: North American Gamma Knife Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12105/12-02
Record Dates: First submitted 2013-03-13; First posted 2013-04-01 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Brain Metastases
Keywords: 1 to 10 measurable brain metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Radiosurgery (SRS) (Experimental): Stereotactic radiosurgery technique via Gamma Knife® Perfexion™ radiosurgical system
  Interventions: Other: Stereotactic radiosurgery (SRS)

INTERVENTIONS:
Other: Stereotactic radiosurgery (SRS) — Dose & prescription The dose will be prescribed to the isodose surface, which encompasses the margin of the metastasis (50-90% [maximum=100%]), as defined by target delineation on the imaging studies.
  The prescribed dose is dependent on the prescription isodose volume (IDV). The prescription IDV is defined as the volume (cm3) that is encompassed by the prescription isodose line (IDL).
  Other Names: Gamma Knife® Perfexion™ radiosurgical system

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, stereotactic radiosurgery (Gamma knife) has on brain metastasis(es). Gamma knife radiosurgery is a way of giving radiation therapy to the brain in a very focused way, so that nearby parts of the brain receive very little exposure to radiation. No incisions are involved. Imaging technology is used to pinpoint the location of the tumor.

In this study, the investigators are also trying to find out how the tumor and/or treatment affect brain function over time. The investigators will do this by performing a series of neurocognitive assessments, or tests of memory, reasoning, and higher brain function, before treatment and at regular intervals after treatment.

DETAILED DESCRIPTION:
This will be a prospective, multi-institution, non-randomized trial of neurocognitive outcomes in patients with multiple, newly-diagnosed brain metastases managed primarily with stereotactic radiosurgery (SRS), specifically the Gamma Knife (GK) system. The goal of the study is to enroll 45 patients with 1-10 newly-diagnosed brain metastases from varied primary cancers with the largest intracranial tumor volume ≤10 cc, ≤15 cc total tumor volume, absence of leptomeningeal disease on MRI, and Karnofsky performance status (KPS) score ≥70 (unless due to intracranial disease), and KPS expected to improve to ≥70 with treatment. The enrolled patients are expected to have fairly good pre-treatment cognitive function, defined as online neurocognitive function (oNCF) assessment scores ≥70 (within 2 standard deviations of mean, 100).

All study participants will undergo standard, pre-treatment clinical evaluations that include: complete clinical/neurologic exam, performance status assessment, systemic staging, and diagnostic MRI of the brain. Upon enrollment, the patients will further undergo high-resolution MRI, including track density imaging (TDI). The baseline neurocognitive function (NCF) will be assessed by a short (20-30 minute) online test battery that can be completed by patients at home, CogState assessment (22 minutes), as well as by a comprehensive neuropsychological evaluation (2-3 hours). The eligible patients will subsequently go on to receive a radiosurgical treatment for their brain metastases.

All patients will have treatment response assessments every 10-12 weeks consisting of a clinical/neurologic exam, performance status evaluation, disease re-staging (if indicated), and diagnostic MRI of the brain. If progressive disease is identified (radiographic progression of treated lesions or new brain lesions), the patients will be considered for "salvage" therapy which will include repeat SRS, whole-brain radiation therapy (WBRT), surgery with or without brachytherapy or best supportive care (e.g. steroids only). The preferred salvage therapy will be SRS provided that the re-treatment criteria are met. Along with regular clinical MRIs, TDI will be obtained.

Mandatory comprehensive follow-up testing by a neuropsychologist (1-2 hours) will occur every 10-12 weeks, starting 4 weeks after completion of SRS, and will continue at these intervals even if salvage therapy is administered for intracranial recurrence. Online NCF testing (oNCF and CogState) will take place in the office setting on the same day as a comprehensive cognitive assessment. Patients will also have the option to do web-based oNCF assessments from home but not more frequently than every 2 weeks. These optional assessments will not be included in the data analysis. All study participants will be followed until death or withdrawal from the study.

The primary aim of the study is to validate the oNCF battery and to demonstrate the feasibility of its use in patients with metastatic brain disease. The former will be accomplished by correlating the findings of the oNCF testing with those of a comprehensive neurocognitive function (cNCF) assessment of a neuropsychologist. Every attempt will be made to identify imaging correlates of neurocognitive function derived from high-resolution MRI, and TDI. The aggregate data in combination with lesion location information (and the corresponding treatment) should provide unique insights into mechanisms that underlie radiation therapy (RT)-related brain injury. Because salvage therapy with WBRT is also permitted and will likely be necessary in a subset of patients, some insights may also be gained on the relative extent, specificity, and temporal evolution of post-treatment NCF dysfunction of each treatment modality.

The data gained from this pilot study could form the basis of future trials of NCF outcomes in cancer patients, especially if oNCF test battery is validated as this may provide a cost-effective method for including NCF outcomes in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of a non-hematopoietic malignancy other than small cell lung cancer and germ cell malignancy within 5 years of registration. If the original histologic proof of malignancy is greater than 5 years, then pathological confirmation is required (e.g. from extra- or intracranial disease).
* Patients with 1-10 measurable brain metastases on a diagnostic-quality contrast-enhanced magnetic resonance imaging (MRI) scan obtained within 30 days prior to registration.
* Patients with ≤10 cc largest tumor volume, and ≤15 cc total tumor volume.
* History/physical examination within 30 days prior to registration.
* If an open biopsy is performed, the patient must be at least one week post biopsy. This requirement does not apply to patients who undergo stereotactic biopsies.
* Age ≥18 years.
* Karnofsky performance status ≥70 (RTOG recursive partitioning analysis (RPA) Class I & II).
* Minimum pre-treatment oNCF score ≥70.
* Patients must provide study-specific informed consent prior to study entry.
* Women of child-bearing age must have a negative, quantitative serum pregnancy test ≤14 days prior to study entry, or have a documented reason why such a test is not necessary (e.g. history of tubal ligation).
* Patients must be able to speak and read English fluently (required for the use of online NCF testing).

Exclusion Criteria:

* Clinical (e.g. multiple cranial nerve deficits in the absence of obvious radiographic disease to explain symptoms) or radiographic evidence of leptomeningeal disease.
* Patients with measurable brain metastasis(es) resulting from small cell lung cancer and/or germ cell malignancy
* No documentation of prior cytotoxic or other therapy for malignancy if such therapy was previously received. Note: This does not apply to patients with synchronous metastases at initial diagnosis.
* Contraindication to MR imaging, such as implanted metal devices or foreign bodies, severe claustrophobia, or contraindications to contrast agent administration.
* Estimated glomerular filtration rate (eGFR) <60 within 6 weeks prior to registration.
* Prior radiation therapy to the brain.
* Severe, active co-morbidity, defined as follows:

  * Unstable angina, and/or congestive heart failure requiring hospitalization within the last 6 months.
  * Transmural myocardial infarction within the last 6 months.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization, or precluding study therapy at the time of registration.
  * Uncontrolled, clinically significant cardiac arrhythmias.
  * Radiologic or clinical evidence of hydrocephalus, or history of previously treated hydrocephalus.
* Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study is potentially teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10-22 (Actual); Study Completion 2015-10-22 (Actual)

PRIMARY OUTCOMES:
Gamma knife radiosurgery treatment | Baseline and 6-months following treatment
  Two short oNCF assessments will be performed at least 30 minutes prior to a clinical neurocognitive function (cNCF) assessments directed by a neuropsychologist at baseline and 6 months following Gamma knife treatment to assess changes in the participants' ability to complete all assessments.
Validation: To estimate consistency in change in z-scores for online oNCF and comprehensive clinical neurocognitive function (cNCF) neurocognitive assessments at baseline and 6-months in the office/clinic setting. | baseline and 6-months following radiosurgery
  * Neuro psychologist will perform assessments: global cognitive function (Montreal Cognitive Assessment (MoCA), fine motor skills (Grooved Pegboard), information processing speed (DKEFS Trails, Symbol-Digit Modality Test), auditory and visual attention (NAB Digit Span, Numbers and Letters A), verbal memory (NAB List Learning and Story Learning), visual memory (NAB Shape Learning and Rey-Osterrieth Complex Figure (ROCF), Brief Visuospatial Memory Test-Revised (BVMT-R™), language (Boston Naming Test, Letter Fluency, Category Fluency, Sentence Repetition), visual-spatial (NAB Visual Discrimination, ROCF) and DKEFS Trails, DKEFS Design Fluency).
  * Patient will complete Quality of Life Questionnaire- Core 30 (QOL-30), Brain Cancer Module-20 (BCM20), and EuroQol Group Questionnaire-5D (EQ-5D) QoL measurements.
  * Patient will complete self-reported measures of depression (BDI-II), anxiety (BAI), qualify of life (FACT-Br), cognition (FACT-COG), and fatigue (Fatigue Severity Scale).

SECONDARY OUTCOMES:
-Feasibility: To demonstrate that at least 95% of participants will have no change from baseline and 12 months after treatment in their ability to complete the online neurocognitive function (oNCF) assessment. | baseline and 12-months after therapy.
  Two short online neurocognitive (oNCF) assessments will be performed. All patients will be required to complete oNCF testing at least 30 minutes prior to a clinical neurocognitive function (cNCF) assessment directed by a neuropsychologist.
- Validation: To estimate consistency and change in scores for online neurocognitive (oNCF) and comprehensive clinical neurocognitive function (cNCF) assessments over all study time points. | baseline and 12-months after treatment.
  To estimate consistency in change in scores for oNCF and cNCF assessments at all study time points. This assessment of change over time can be achieved by employing an analysis of covariance model that relates the continuous assessment outcome to the classification factor (oNCF or cNCF) and the continuous covariate, time of neurocognitive exam, as well as an interaction term. Estimates of zero for the interaction term and classification factor will indicate consistency.

OTHER OUTCOMES:
To determine what healthcare cost data can be collected in patients with metastatic disease with the aim of estimating the relative healthcare cost of the Gamma Knife radiosurgery (prospective cost data collection). | Participants will be followed for the duration of hospital stay and initial follow up, an expected average of 6 weeks
  The billing data will be obtained from radiation oncology, neurosurgery, and hospital billing departments during the trial period every quarter. A 'Medicare' costing approach will convert hospital charges to costs, using publicly available information from Medicare cost reports. Charges will not be reported publicly. Proprietary costs accounting information will not be requested. The purpose of this data collection is to determine what data can be collected in patients with metastatic disease within a context of a multi-institutional trial. Since this approach has not previously been done in a context of a prospective, multi-institutional clinical trial in a patient population with metastatic disease, any post hoc analysis will be subject to the availability of the collected data but every attempt will be made to determine direct and indirect costs of the study treatments.
Document the incidence of asymptomatic and symptomatic radiation necrosis in patients treated with gamma knife radiosurgery with or without whole brain radiation therapy WBRT (if WBRT is offered as salvage therapy) | 12 months post radiosugery
  Percentage of patients who experience asymptomatic and symptomatic radiation necrosis will be provided in frequency tables

CONTACTS AND LOCATIONS:
Overall Officials: Igor J Barani, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States